CLINICAL TRIAL: NCT06259331
Title: Evaluation of the Excretion of Viloxazine and Its Metabolite 5-Hydroxy-viloxazine Glucuronide Into Breast Milk Following Multiple Doses of SPN-812 (600mg, QD) in Healthy Lactating Women
Brief Title: Evaluation of Viloxazine and Its Metabolite 5-Hydroxy-viloxazine Glucuronide Into Breast Milk in Healthy Lactating Women
Acronym: SPN-812
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 812P418
Record Dates: First submitted 2024-01-17; First posted 2024-02-14 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Healthy Lactating Women
Keywords: Healthy Lactating Women; Healthy Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): Up to 15 healthy, lactating women will be enrolled in the study.
  Interventions: Drug: SPN-812 (600mg, QD)

INTERVENTIONS:
Drug: SPN-812 (600mg, QD) — Viloxazine ER

SUMMARY:
This is an open label, single treatment, multiple doses lactation study of SPN-812 in healthy lactating women. The study is designed to assess the excretion of viloxazine and its major metabolite 5-HVLX-gluc into breast milk following repeated administration of SPN-812 600 mg, QD.

This study is comprised of Screening, Inpatient Admission, Treatment Period and End of Study (EOS). The total duration of the study is up to 32 days including Screening up to 28 days and 4 days of Treatment Period. Subjects will remain in the inpatient unit for 5 days, including the day of admission to the inpatient unit (Day -1), 3 days of dosing SM (Days 1-3), and the day of discharge (Day 4).

DETAILED DESCRIPTION:
This is an open label, single treatment, multiple doses, lactation study of SPN-812 at steady state in healthy lactating women. The study is designed to assess the excretion of viloxazine and its major metabolite 5-HVLX-gluc into breast milk following repeated administration of SPN-812 600 mg daily for 3 days. The study is designed to assess the excretion of viloxazine and its major metabolite 5-HVLX-gluc into breast milk following repeated administration of SPN-812 600 mg, QD.

This study is comprised of Screening, Inpatient Admission, Treatment Period, End of Study (EOS) with FU phone call. The total duration of the study is up to 32 days including Screening up to 28 days and 4 days of Treatment Period. Subjects will remain in the inpatient unit for 5 days, including the day of admission to the inpatient unit (Day -1), 3 days of dosing SM (Days 1-3), and the day of discharge (Day 4).

Subjects will complete the screening visit, after informed consent is obtained, within 28 days prior to dose initiation. Inclusion/exclusion criteria will be reviewed to determine the subject's eligibility at Screening. A lactation consultant will be available to provide lactation support to subjects once they are enrolled.

Since the mother's infant cannot receive breast milk for 7 consecutive days (Day-1 to Day 6), the mother will be reminded at Screening to make plans to have their infant fed 7 consecutive days with either (a) formula or (b) stored breast milk (e.g., breast milk pumped and stored in the freezer during the screening period between the screening visit and the day of admission to inpatient unit).

Subjects will be admitted to the inpatient unit on Day -1 to confirm eligibility. Subjects will receive 600 mg SPN-812 in the morning of Days 1, 2 and 3 after completion of safety assessments. SM should be administered at the same time in the morning (±30 min) of dosing days. Breast milk and blood sample for PK analysis will then be collected on Day 3 per schedule. Non-PK breast milk expressed on Days -1, 1, and 2 will be collected over the time intervals and these samples will not be analyzed for drug concentrations. The volume and the start and end times of the collection of each non-PK and PK breast milk sample will be recorded. The end of study (EOS) procedures will be conducted prior to discharge on Day 4 following the last breast milk and blood sample collection. If subject discontinues early, all EOS procedures will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy lactating females, 18 to 45 years of age, who are actively breastfeeding (including baby to breast, bottle feeding mother's expressed breast milk) and are at least 12 weeks postpartum of a healthy term newborn infant (no medical complications) and not more than 2 years postpartum. Lactation must be well established and the mother is exclusively breast feeding her baby (not providing supplemental formula) prior to the day of admission to inpatient unit.
2. Has a body mass index between 18 to 35 kg/m2, included.
3. Is considered medically healthy by the Investigator via assessment of physical examination (neurological examinations included), medical history, clinical laboratory tests, vital signs, Columbia-Suicide Severity Rating Scale (C-SSRS) and electrocardiogram (ECG).
4. Is willing to temporarily discontinue breastfeeding their infant and discard all their breast milk for 7 consecutive days, including day of admission to inpatient unit (Day -1), 3 consecutive days of dosing SM while in the inpatient unit (Days 1 to 3), and 3 consecutive days after last dose of SM (including day of discharge from the inpatient unit and 2 days at home; Days 4 to 6); and willing to store sufficient amount of breast milk (e.g., breast milk pumped and stored in freezer before the day of admission), and/or infant formula to feed infant during these 7 consecutive days.
5. Is either sexually inactive (abstinent) or, if sexually active, must agree to use/practice one of the following acceptable birth control methods beginning during the screening period prior to the first dose of SM, throughout the inpatient study, and for 3 days following the last dose of SM (Day 3):

   * intra-uterine contraceptive device;
   * barrier method: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository;
   * is surgically sterile or male partner is surgically sterile;
   * established use of a patch, vaginal ring, oral, injected or implanted hormonal methods of contraception that can be used in lactating women;
   * Essure® procedure performed at least 6 months prior to Screening and had hysterosalpingogram after the Essure procedure to document tubal occlusion prior to screening.
6. Must not be in the process of weaning before admission and have maintained an adequate breast milk supply with regularly pumping or routine breastfeeding (e.g., pumping or feeding 3-4 times a day) at admission.
7. Is currently a non-smoker who has not used tobacco or nicotine-containing products (chewed or smoked) or replacement products, including electronic cigarettes, within 3 months prior to screening and a negative cotinine test result at Screening.
8. Agrees to use only the emollient or nipple cream recommended by the investigator for use during the sampling period, if needed.
9. Able to voluntarily provide written informed consent to participate in the study.
10. Able to understand and willing to comply with all study requirements.
11. Able and willing to swallow capsules whole, without crushing, chewing, or cutting.

Exclusion Criteria:

1. Participation in any other investigational study drug trial in which receipt of an investigational study drug within 30 days or 5 half-lives before Screening, whichever is longer.
2. Is unwilling or unable to comply with the Lifestyle guidelines presented in the protocol during the study period.
3. Has history or presence of clinically significant systemic disease (including psychological and psychiatric disorders).
4. Is currently using, or tests positive at Screening for cotinine, alcohol, or drugs (opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates, PCP, benzodiazepines, and THC/cannabis).
5. Is pregnant (has positive serum pregnancy test at Screening) or becomes pregnant during study (has positive urine pregnancy test).
6. Has history of breast implants, breast augmentation, or breast reduction surgery.
7. Has history of mastitis within 30 days, breast cancer and/or has had a mastectomy or lumpectomy with the exception of a benign fibroma or lipoma removal at the investigator's discretion; and/or a clinically significant abnormality observed in either breast during a clinical breast exam at Screening or Admission (Day -1).
8. Has a history of alcohol use disorder within 1 year of Screening; or assessed by the PI as having regularly consumed alcohol exceeding 14 units per week (1 unit equals 340 mL of beer, 115 mL of wine, or 43 mL of spirits) within 1 year of Screening.
9. Is using recreational or illicit drug(s) (e.g., cannabis /tetrahydrocannabinol (THC), opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates, and benzodiazepines) within 1 year of Screening.
10. Has clinically significant vital signs abnormalities (systolic blood pressure less than 90 or greater than 140 mmHg, diastolic blood pressure less than 60 or greater than 90 mmHg, or pulse rate (PR) less than 50 or greater than 100 bpm at Screening.
11. Has a clinical laboratory test values outside the reference range at Screening that, in the opinion of the investigator, are clinically significant, or any of the following:

    * Serum creatinine >1.5 times the upper limit of normal (ULN)
    * Serum total bilirubin >1.5 times ULN
    * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times ULN
12. Has clinically significant ECG abnormalities at Screening, including:

    * PR interval >220 ms
    * QRS interval >130 ms
    * QTcF interval >470 ms
13. Has any disease or medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability, or interfere with the conduct or interpretation of the study.
14. Has evidence of infection with hepatitis B and C, and human immunodeficiency virus HIV-1 and HIV-2, as determined by results of testing at Screening.
15. Has a condition or planned procedure that may interfere with the absorption, metabolism, or elimination of the study drug (e.g., cholecystectomy).
16. Is using prescription medication within 14 days prior to administration of SM or 5 half-lives, whichever is longer, with the exception of hormonal contraceptives.
17. Is using over-the-counter products (including vitamins, herbal products and natural food supplements) within 14 days prior to administration of SM or 5 half-lives, whichever is longer. Exceptions include postnatal vitamins, topical products without systemic absorption and acetaminophen (< 2 g/day).
18. Has an allergy to viloxazine.
19. Has an Edinburgh Postnatal Depression Scale score >13.
20. Has attempted suicide within the 6 months prior to Screening or is at significant risk of suicide (either in the opinion of the Investigator or defined as a "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the 12 months prior to screening).
21. In the investigator's opinion, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cai, Study Director — Clinical Pharmacology; Darin B Brimhall, DO, Principal Investigator — PPD Phase I Clinic
Locations (1):
- PPD Phase I Clinic, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Up to 15 healthy, lactating women will be enrolled in the study.
  SPN-812 (600mg, QD): SPN-812 (600mg, QD)
Period: Overall Study
Arm/Group | Cohort 1
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Up to 15 healthy, lactating women will be enrolled in the study.
  SPN-812 (600mg, QD):
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (4.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Pre-dose Viloxazine Concentrations in Plasma [Mean (Standard Deviation); unit: µg/mL] | 0.0 (0.0)
Pre-dose Metabolite Concentrations in Plasma [Mean (Standard Deviation); unit: µg/mL] | 0.0 (0.0)
Pre-dose Viloxazine concentration in Breast milk [Median (Standard Deviation); unit: µg/mL] | 0.0 (0.0)
Pre-dose Metabolite concentration in Breast Milk [Mean (Standard Deviation); unit: µg/mL] | 0.0 (0.0)

OUTCOME MEASURES:

1. Primary Outcome: AUCtau,Milk
Description: Area under the concentration-time curve over a 24-hour dosing interval in breast milk for viloxazine and its metabolite 5-HVLX-gluc
Time Frame: Day 3: -4 to <0 hours pre-dose, and '0 to 4', '4 to 6', '6 to 8', '8 to 10', '10 to 12', '12 to 16' and '16 to 24' hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•h/mL, (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg•h/mL, (CV%)
  Viloxazine | 21.4 (34.4)
  5-HVLX-gluc | 1.59 (31.1)

2. Primary Outcome: Cmax,Milk
Description: Maximum observed concentration in breast milk for viloxazine and its metabolite 5-HVLX-gluc
Time Frame: -4 to <0 hours pre-dose, and '0 to 4', '4 to 6', '6 to 8', '8 to 10', '10 to 12', '12 to 16' and '16 to 24' hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL, (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg/mL, (CV%)
  Viloxazine | 1.41 (33.1)
  5-HVLX-gluc | 0.0940 (31.1)

3. Primary Outcome: Tmax,Milk
Description: time of maximum observed concentration in breast milk for viloxazine and its metabolite 5-HVLX-gluc
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h (min to max)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
h (min to max)
  Viloxazine | 5.53 [3.54 to 7.60]
  5-HVLX-gluc | 9.53 [5.63 to 15.59]

4. Primary Outcome: Ctrough,Milk
Description: Observed drug concentration in milk immediately before the next dose for viloxazine and its metabolite 5-HVLX-gluc
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg/mL (CV%)
  Viloxazine | 0.426 (48.4)
  5-HVLX-gluc | 0.0480 (33.3)

5. Primary Outcome: Cave,Milk
Description: Average drug concentration in milk, calculated as the ratio of AUCtau,milk/24 for viloxazine and its metabolite 5-HVLX-gluc
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg/mL (CV%)
  Viloxazine | 0.912 (34.3)
  5-HVLX-gluc | 0.0677 (30.7)

6. Secondary Outcome: Plasma AUCtau,ss
Description: Area under the concentration-time curve over the dosing interval (AUCtau) in plasma for viloxazine and its metabolite 5-HVLX-gluc at steady-state
Time Frame: Day 3 pre-dose, and Day 3 at 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 16.0 and 24.0-hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•h/mL, (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg•h/mL, (CV%)
  Viloxazine | 63.4 (28.2)
  5-HVLX-gluc | 42.3 (21.0)

7. Secondary Outcome: Plasma Cmax,ss,
Description: Maximum observed concentration in plasma for viloxazine and its metabolite 5-HVLX-gluc
Time Frame: Day 3 pre-dose, and Day 3 at 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 16.0 and 24.0-hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL, (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg/mL, (CV%)
  Viloxazine | 3.92 (23.7)
  5-HVLX-gluc | 2.73 (19.3)

8. Secondary Outcome: Plasma Tmax,ss
Description: Time to Peak Concentration
Time Frame: Day 3 pre-dose, and Day 3 at 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 16.0 and 24.0-hours post-dose.
Measure: Median (Full Range); unit: h (min to max)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
h (min to max)
  Viloxazine | 5.00 [0.50 to 6.03]
  5-HVLX-gluc | 6.00 [5.00 to 8.00]

9. Secondary Outcome: Plasma CL/Fss,
Description: Apparent clearance (Dose/AUCtau,ss)
Time Frame: Day 3 pre-dose, and Day 3 at 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 16.0 and 24.0-hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h, (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
L/h, (CV%)
  Viloxazine | 9.46 (28.2)
  5-HVLX-gluc | NA (NA) — Not Calculated. From the mass balance study, it was identified that the major metabolite of viloxazine following oral SPN-812 (viloxazine) was 5-HVLX-gluc; however, the factor of in vivo conversion of viloxazine to 5-HVLX-gluc is not known. Therefore, the amount of 5-HVLX-gluc to estimate total clearance of 5-HVLX-gluc, i.e., the amount in equation to calculate the CL/Fss = (Amount of 5-HVLX-gluc/AUC of 5-HVLX-gluc) is not known and the CLss/F of 5-HVLX-gluc is not calculable.

10. Secondary Outcome: Plasma Cave,ss
Description: Average plasma concentration, calculated as the ratio of AUCtau,ss/24
Time Frame: Day 3 pre-dose, and Day 3 at 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 16.0 and 24.0-hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL, (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg/mL, (CV%)
  Viloxazine | 2.64 (28.3)
  5-HLVX-gluc | 1.76 (21.0)

11. Secondary Outcome: Plasma Ctrough,ss
Description: Observed plasma concentration immediately before the next dose
Time Frame: Day 3 pre-dose, and Day 3 at 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 16.0 and 24.0-hours post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL, (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
µg/mL, (CV%)
  Viloxazine | 1.36 (46.7)
  5-HVLX-gluc | 0.878 (27.3)

12. Secondary Outcome: Breast Milk-plasma Ratio (ML/PL)
Description: Breast milk-plasma ratio (ML/PL) based on AUC over 24 hours for viloxazine and 5-HVLX-gluc at plasma steady-state. Ratio of AUCtau from milk to AUCtau from plasma (CV%)
Time Frame: Breast Milk PK Day 3: -4 to <0 hrs pre-dose, and '0 to 4', '4 to 6', '6 to 8', '8 to 10', '10 to 12', '12 to 16' and '16 to 24' hrs post-dose, Plasma PK Day 3 pre-dose, and Day 3 at 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 16.0 and 24.0-hrs post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
Ratio (CV%)
  Viloxazine | 0.338 (17.4)
  5-HVLX-gluc | 0.0376 (28.4)

13. Secondary Outcome: Estimated Daily Infant Dosage (EDID, mg/kg/Day)
Description: Estimated daily infant dosage (mg/kg/day) calculated as Milk/Plasma Ratio x the average maternal plasma concentration (Cave,ss) multiplied by 150 mL/kg/day (EDID 150) and 200 mL/kg/day (EDID 200), respectively.
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/kg/Day (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
mg/kg/Day (CV%)
  Viloxazine EDID 150 | 0.134 (34.4)
  5-HVLX-gluc EDID 150 | 0.00994 (31.1)
  Viloxazine EDID 200 | 0.178 (34.4)
  5-HVLX-gluc EDID 200 | 0.0133 (31.1)

14. Secondary Outcome: Relative Infant Dose (RID, %) at Plasma Steady-state
Description: Relative infant dose (%); the percent of the weight-adjusted maternal dosage consumed in breast milk over 24 hours, calculated as EDID (mg/kg/day)/maternal dosage (mg/kg/day) multiplied by 100 %.
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
Percent (CV%)
  Viloxazine RID 150 (%) (based on EDID 150) | 1.53 (27.6)
  5-HVLX-gluc 150 (%) (based on EDID 150) | 0.114 (38.2)
  Viloxazine RID 200 (%) (based on EDID 200) | 2.04 (27.6)
  5-HVLX-gluc 200 (%) (based on EDID 200) | 0.152 (38.2)

15. Secondary Outcome: Daily Infant Dosage (DID)
Description: Daily infant dosage (mg/day); total drug present in breast milk and consumed by the infant per day, which is equal to AM,milk.
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/day (CV%)
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
mg/day (CV%)
  Viloxazine | 0.511 (69.8)
  5-HVLX-gluc | 0.0357 (48.2)

16. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: All subjects who are enrolled and who receive SM will be monitored and questioned regarding the occurrence of AEs. Adverse events occurring prior to SM administration on Study Day 1 will become part of the subject's medical history. Throughout the study, the Investigator must seek information on AEs by specific questioning and, as appropriate, by examination.
Time Frame: 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 15
Participants | 12

ADVERSE EVENTS:
Time Frame: 11 days
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 12/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=15)
somnolence (Nervous system disorders) | 10 (10)
dizziness (Nervous system disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 3 (3)
breast tenderness (Reproductive system and breast disorders) | 3 (3)
headache (Nervous system disorders) | 2 (2)
dry mouth (Gastrointestinal disorders) | 2 (2)
decreased appetite (Metabolism and nutrition disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1)
chills (General disorders) | 1 (1)
dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT06259331/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT06259331/SAP_001.pdf